CLINICAL TRIAL: NCT01715012
Title: A Phase 2a Randomized, Double Blind, Placebo Controlled, Single-center Study of ST266 Spray in Diabetic Subjects With Deep Burns Managed With Meshed Skin Grafts.
Brief Title: Study of ST266 in Diabetic Subjects With Deep Burns Managed With Skin Grafts
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Enrollment futility
Sponsor: Noveome Biotherapeutics, formerly Stemnion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ST-03-12
Record Dates: First submitted 2012-10-22; First posted 2012-10-26 (Estimated); Last update posted 2019-05-15 (Actual); Status verified 2019-05

CONDITIONS: Third Degree Burns; Diabetes
Keywords: Burn; Diabetes; Skin graft; Donor site
MeSH Terms: conditions — Diabetes Mellitus; Burns | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ST266 (Experimental): ST266 sprayed to the skin graft and donor site
  Interventions: Biological: ST266
- Saline (Placebo Comparator): Saline (placebo)sprayed to the skin graft and donor site
  Interventions: Drug: Saline

INTERVENTIONS:
Biological: ST266 — ST266 is applied daily by spray to burn wound and skin graft donor site
  Arms: ST266
Drug: Saline — Saline is applied daily by spray to burn wound and skin graft donor site
  Other Names: Placebo
  Arms: Saline

SUMMARY:
This study is a randomized, double blind, placebo controlled trial at a single site. The primary objective is to evaluate the safety of ST266 in diabetic subjects with deep burns. The secondary objectives of this study are to (1) evaluate efficacy of ST266 in healing burns and (2) evaluate whether treatment with ST266 results in less scarring, in subjects with diabetes separately comparing healing of the skin graft and the skin graft donor site using ST266 plus a burn dressing versus placebo and a burn dressing.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated Institutional Review Board-approved written Informed Consent
* 18 - 75 years of age.
* Thermal or scald burn, either full thickness or deep partial thickness, which in the opinion of the burn surgeon, requires a meshed skin graft to heal.
* Target burn area for treatment equal to or less than three percent total body surface area.
* A skin graft site harvested at 10/1000ths of an inch and a skin graft meshed at 2:1.
* Total Body Surface Area (TBSA) burn of less than or equal to 20 percent total body surface.
* Patient must have a known history of diabetes, or be found to have diabetes at the time of admission, confirmed by a Hemoglobin A1C of greater than 6.5 percent.
* If a woman of child-bearing potential (WOCBP), she and her partner must be willing to employ either a highly effective form of birth control (e.g., implants, injectable medications, a hormone combination oral contraceptive, etc.), sexual abstinence, or a vasectomised partner, in combination with a barrier method, for the entire duration of the study (through study discharge). Male subjects with a WOCBP partner must be willing to use a condom during sexual activity for the entire duration of the study (through study discharge).
* Willing to participate in the clinical study and comply with the requirements of the trial.

Exclusion Criteria:

* Full thickness burns involving tendon, ligament, bone, or joint capsule.
* Burns of the face, neck, palmer surface of the hands and plantar surface of the foot.
* Burn from chemical, electrical or radiation causes.
* Subjects with any immune deficiency including current treatment with corticosteroid medication, chemotherapeutic agents, anti-viral therapy, or concurrent radiation therapy within 30 days of signing the informed consent.
* Active cancer or a history of cancer in the five years prior to signing the informed consent form. (History of basal cell carcinoma is allowed).
* Life expectancy of less than one year.
* Patients requiring care in the Intensive Care Unit.
* Inhalation injury requiring mechanical ventilation.
* Multiple trauma (significant traumatic injury to a solid organ in addition to skin).
* Psychiatric condition or substance abuse which in the Investigator's opinion may pose a threat to subject compliance.
* History of non-compliance with treatment or clinical visit attendance.
* Participation in an investigational trial within 30 days of study entry.
* Women who are pregnant or lactating
* Prisoners
* Acute clinically significant infection (including viral infections) in the six weeks prior to administration of study drug or any clinically significant ongoing chronic infection (excluding fungal infections of the nail beds).
* Evidence or history of skin conditions that would interfere with evaluations.
* Any other uncontrolled concomitant disease, condition, or treatment that could interfere with the conduct of the study, or that would, in the opinion of the investigator, pose an unacceptable risk to individuals in this study or interfere with the interpretation of study data.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2012-10; Primary Completion 2015-01 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Safety | Beginning at enrollment and continuing 12 months after last treatment
  The primary objective of this study is to evaluate the safety of ST266 in treating burns in diabetic subjects by evaluating adverse events and serious adverse events. Physical examination, hematology, serum chemistry, urinalysis, vital signs, Adverse Event monitoring, and concomitant medications, cytokine and antibody levels will be monitored at baseline and during the study.

SECONDARY OUTCOMES:
Healing of skin graft | Up to 2 weeks of treatment
  Evaluation of ST266 compared with placebo (saline) in treating burns in diabetic subjects by assessing the time to complete healing of the skin graft.
Healing of skin graft donor site | Up to 2 weeks of treatment
  Evaluation of ST266 compared with placebo (saline) in treating burns in diabetic subjects by assessing the healing of the skin graft donor site.
Scarring of skin graft | One year following treatment
  Evaluation of ST266 compared with placebo (saline) in treating burns in diabetic subjects by assessing scarring of the skin graft at six months and one year using a validated scar scale.
Scarring of skin graft donor site | One year following treatment
  Evaluation of ST266 compared with placebo (saline) in treating burns in diabetic subjects by assessing scarring of the skin graft donor site at six months and one year using a validated scar scale.

CONTACTS AND LOCATIONS:
Overall Officials: Larry Jones, MD, Principal Investigator — Ohio State University
Locations (1):
- The Burn Unit of the Wexner Medical Center at The Ohio State University., Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No